CLINICAL TRIAL: NCT04287361
Title: Efficacy of Intravenous Clonazepam According to the Dosage in Children Status Epilepticus
Brief Title: Clonazepam in Children Status Epilepticus
Acronym: UHAPA
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0501
Record Dates: First submitted 2020-02-11; First posted 2020-02-27 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Epilepticus Status
MeSH Terms: conditions — Status Epilepticus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Loading dose < 0,03 mg/kg: Patient being treated for a status epilepticus who received an initial dose of clonazepam < 0.03 mg / kg
  Interventions: Other: Efficacy of intravenous clonazepam
- Loading dose ≥ 0,03 mg/kg: Patient being treated for a status epilepticus who received an initial dose of clonazepam ≥ 0.03 mg / kg
  Interventions: Other: Efficacy of intravenous clonazepam

INTERVENTIONS:
Other: Efficacy of intravenous clonazepam — Efficacy of intravenous clonazepam

SUMMARY:
•Background: Intravenous clonazepam is the most widely used first-line benzodiazepine in Europe for the initial management of status epilepticus in children.

The guidelines of the "Société de reanimation de langue francaise" (SRLF) and the "société française de médecine d'urgence" (SFMU) published in 2018 recommend an initial loading dose of 0.015 mg / kg of clonazepam in this situation (maximum 1.5 mg).

To our knowledge, there is no specific study of the efficacy of clonazepam according to the dose used.

Objective: To compare the effectiveness of the initial loading dose of clonazepam in children treated for status epilepticus

•Methods: Monocentric retrospective study including children < 16 years who have benefited from an initial loading dose of clonazepam in the context of status epilepticus treated at the Montpellier University Hospital between January 2016 and June 2019.

The investigators collected data from medical records (clinic, treatment , evolution) and compared these according to the dosage of clonazepam used.

•Discussion: Among the benzodiazepines used in the first-line treatment of pediatric status epileptic, lorazepam and midazolam are the most widely used drugs in the world.

Lorazepam is not so much used in Europe because the injectable form is not available for a daily use. Conversely, clonazepam is used in a large number of European countries but is rarely used in the United States due to the lack of an injectable form.

About the tolerance of treatment, except overdose situations, clonazepam is a drug well tolerated in the pediatric populatin. The main side effects of clonazepam are respiratory depression and impaired alertness.

To our knowledge, this study is the first to examine the efficacy depending on the initial loading dosage of clonazepam in children status epilepticus.

ELIGIBILITY:
Inclusion criteria:

An individual must fulfill all of the following criteria in order to be eligible for study enrollment:

* Aged under 16 years
* Status epilepticus taken care of at the CHU de Montpellier

Exclusion criteria

● No loading dose of clonazepam

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: An individual must fulfill all of the following criteria in order to be eligible for study enrollment:
  * Aged under 16 years
  * Status epilepticus taken care of at the CHU de Montpellier
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
effectiveness in stopping seizures | 1 day
  The primary endpoint was clinical cessation of seizures, which was defined as the absence of clinical signs of seizures immediately following the injection of clonazepam.

SECONDARY OUTCOMES:
need for a second dose of clonazepam | 1 day
  need for a second dose of clonazepam
duration of seizure | 1 day
  duration of seizure (minutes)
type of seizures | 1 day
  type of seizures (focal, generalized);
aetiologies ; | 1 day
  aetiologies (idiopathic, symptomatic)
pre-hospital treatment used | 1 day
  pre-hospital treatment used
whether or not to use a dose greater than one milligram | 1 day
  whether or not to use a dose greater than one milligram
introduction of a maintenance dose | 1 day
  introduction of a maintenance dose
using another antiepileptic drug | 1 day
  using another antiepileptic drug (phenobarbital, fosphenytoin, thiopental)
Hospitalization in an intensive care or resuscitation unit | 1 day
  Hospitalization in an intensive care or resuscitation unit
Rate of hospitalization in conventional sector | 1 day
  Rate of hospitalization in conventional sector
introduction of antiepileptic treatment after treatment | 1 day
  introduction of antiepileptic treatment after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maxime colmard, résident, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC